CLINICAL TRIAL: NCT06474481
Title: A Study of the Zanubrutinib With G-CHOP Regimens in the Frontline Treatment of Intermediate-high Risk Follicular Lymphoma
Brief Title: Zanubrutinib and G-CHOP in Untreated Intermediate-high Risk Follicular Lymphoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TN-FL001
Record Dates: First submitted 2024-06-12; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: FL
Keywords: Zanubrutinib; Intermediate-high risk Follicular Lymphoma; G-CHOP
MeSH Terms: interventions — zanubrutinib; obinutuzumab; Prednisone; Cyclophosphamide; Vincristine; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental): Induction: Zanubrutinib and G-CHOP 4-6cycles
  Maintenance: Zanubrutinib and Obinutuzumab 1 year
  Interventions: Drug: Zanubrutinib; Drug: Obinutuzumab; Drug: Prednisone; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Doxorubicin

INTERVENTIONS:
Drug: Zanubrutinib — Zanubrutinib, 160mg PO BID.on days 1-28 Induction treatment: 4-6cycles ; Maintenance: 1 year;
Drug: Obinutuzumab — Induction treatment: Obinutuzumab (G), 1000mg, IV, D1/8/15 (C1), D1 (C2-4/6); for 4-6 cycles, 1 cycle = 28 days Maintenance: Obinutuzumab (G), 1000mg, IV, every 2 months for 1 year;
Drug: Prednisone — Prednisone (P), 100 mg, PO, D2-6；for 4-6 cycles for CHOP treatment , 1 cycle = 28 days
Drug: Cyclophosphamide — Cyclophosphamide (C), 750 mg/m2, IV, D2; for 4-6 cycles for CHOP treatment , 1 cycle = 28 days
Drug: Vincristine — Vincristine (O), 1.4 mg/m2 (maximum 2 mg), IV, D2; for 4-6 cycles for CHOP treatment , 1 cycle = 28 days
Drug: Doxorubicin — Doxorubicin (H), 50 mg/m2, IV, D2; for 4-6 cycles for CHOP treatment ，1 cycle = 28 days

SUMMARY:
:This is a an open-label, single-arm study to evaluate the efficacy and safety of zanubrutinib and G-CHOP in untreated Intermediate-high risk Follicular Lymphoma patients.

ELIGIBILITY:
Inclusion criteria.

1. Histologically confirmed CD20 positive (+) follicular lymphoma, grade 1, 2, or 3a
2. Have had no prior systemic treatment for lymphoma
3. Meeting Groupe d'Etude des Lymphomes Folliculaires (GELF) criteria for initiation of treatment
4. 18-75 years old.
5. ECOG Performance Status of 0-2 within 10 days prior to registration.
6. Stage II, III, or IV by Ann Arbor staging system.
7. defined as Intermediate-high risk by the follicular lymphoma international prognostic index (FLIPI) 1 or FLIPI 2.
8. Demonstrate adequate organ function as defined below; all screening labs to be obtained within 28 days prior to registration.

   * Hematological: WBC≥3.5×109/L, Platelets ≥ 75×109/L,Absolute Neutrophil Count (ANC) ≥ 1.0×109/L，Hemoglobin (Hgb) ≥ 80 g/L
   * Renal:Calculated creatinine clearance ≥ 50 mL/min
   * Hepatic:Bilirubin ≤ 1.5 × upper limit of normal (ULN), AST/ALT ≤ 2.5×ULN
9. Females of childbearing potential must be willing to abstain from vaginal intercourse or use an effective method(s) of contraception from the time of informed consent, during the study and for 6 months after the last dose of study drug(s). Males able to father a child must be willing to abstain from vaginal intercourse or to use an effective method(s) of contraception from initiation of treatment, during the study and for 3 months after the last dose of study drug(s). See the protocol.
10. Life expectancy ≥6 months
11. Sign (or their legally-acceptable representatives must sign) an informed consent document indicating that they understand the purpose of and procedures required for the study, including biomarkers, and are willing to participate in the study

Exclusion criteria:

1. Known active central nervous system lymphoma or leptomeningeal disease
2. Evidence of diffuse large B-cell transformation
3. Grade 3b FL
4. Concurrent malignancy or malignancy within the last 3 years (except for ductal breast cancer in situ, non-melanoma skin cancer, prostate cancer not requiring treatment, and cervical carcinoma in situ) whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen are not eligible for this trial
5. Known history of human immunodeficiency virus (HIV), or active hepatitis C Virus, or active hepatitis B Virus infection, or any uncontrolled active significant infection, including suspected or confirmed John Cunningham (JC) virus infection
6. Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any class 3 (moderate) or class 4 (severe) cardiac disease as defined by the New York Heart Association functional classification. Or left ventricular ejection fraction <50%;
7. Neuropathy ≥grade 2
8. Known history of human immunodeficiency virus (HIV), or active hepatitis C Virus, or active hepatitis B Virus infection, or any uncontrolled active significant infection
9. Known pneumonia associated with idiopathic pulmonary fibrosis, machine (for example, occlusive bronchiolitis), history of drug induced pneumonia, or screening during the chest computed tomography (CT) showed active pneumonia
10. Have serious neurological or psychiatric history, can't normal study, including dementia, epilepsy, severe depression and mania
11. Patients who were deemed by the investigator to be ineligible for enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
CR (complete response) rate after induction (4 or 6 Cycles) by investigator (INV) | From enrollment to the end of treatment at cycle 4 or 6 (each cycle is 28 days)
  Percentage of participants with complete response was determined on the basis of investigator assessments according to 2014 Lugano criteria

SECONDARY OUTCOMES:
Objective Response rate after induction by investigator (INV) | From enrollment to the end of end of treatment at cycle 4 or 6 (each cycle is 28 days)
  ORR is defined as the proportion of patients achieving complete response (CR) or partial response (PR), as determined by INV according to 2014 Lugano criteria
Overall survival (OS) | From the date of cycle 1, day 1 to the date of death regardless of cause, assessed up to 3 years
  Overall survival (OS) is defined as the duration from the date of initiation of the first cycle of treatment to the date of death because of any cause
Progression free survival (PFS) | From the date of cycle 1, day 1 to the date of death regardless of cause, assessed up to 3 years
  -PFS defined as time from the date of enrollment to the date of first confirmed disease progression or death due to any cause, whichever occurs first, as determined by INV

IPD SHARING:
Plan to Share IPD: Undecided